CLINICAL TRIAL: NCT01019473
Title: A Multi-centre, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multiple Oral Dose Titration Proof of Concept Study in Patients With Huntington's Disease to Assess the Efficacy, Safety and Tolerability of AFQ056 in Reducing Chorea
Brief Title: Efficacy, Safety and Tolerability of AFQ056 in Patients With Huntington's Disease in Reducing Chorea
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFQ056A2207; 2009-011743-39
Record Dates: First submitted 2009-11-19; First posted 2009-11-25 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Huntington's Disease; Chorea
Keywords: Huntington's disease; Chorea; Dyskinesia
MeSH Terms: conditions — Huntington Disease; Chorea; Dyskinesias | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AFQ056A (Experimental)
  Interventions: Drug: AFQ056
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056
  Arms: AFQ056A
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will assess the efficacy, safety and tolerability of AFQ056 when added to optimize standard therapy in patients that have Huntington's disease in reducing chorea.

ELIGIBILITY:
Inclusion Criteria:

* Huntington's disease (based on DNA testing polyQ >36) with a UHDRS maximal chorea score of >10
* patient with concomitant Huntington's medication (anti-depressants, neuroleptics, benzodiazepines) are allowed but the total daily dose and dosing regimen has to be stable for at least one months prior to randomization
* female patients without childbearing potential (post-menopausal or surgically sterilized), all patients must using a double-barrier local contraception

Exclusion Criteria:

* patients with marked cognitive impairment (MMSE less than 18), with presence of psychosis and/or confusional states
* patients with a history or presence of renal impairment and/or liver disease Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of AFQ056 on the severity of chorea in Huntington's disease measured by Unified Huntington's Disease Rating Scale (UHDRS) Maximal Chorea score. | Baseline to day 28

SECONDARY OUTCOMES:
Potential effect of AFQ056 on the motor, cognitive, behavioral and functional assessments using UHDRS. | Day 1 to day 46
Potential effect of AFQ056 on functional and quality of life scales, neuropsychiatric assessments and cognitive assessments in Huntington's Disease patients | Day 1 to day 46

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Germany (6):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Bochum
  - Novartis Investigator Site, Münster
  - Novartis Investigator Site, Taufkirchen
  - Novartis Investigator Site, Tübingen
  - Novartis Investigator Site, Ulm
- United Kingdom (4):
  - Novartis Investigator Site, Birmingham
  - Novartis Investigator Site, Cardiff
  - Novartis Investigator Site, Manchester
  - Novartis Investigator Site, Oxford

REFERENCES:
- [Derived] Reilmann R, Rouzade-Dominguez ML, Saft C, Sussmuth SD, Priller J, Rosser A, Rickards H, Schols L, Pezous N, Gasparini F, Johns D, Landwehrmeyer GB, Gomez-Mancilla B. A randomized, placebo-controlled trial of AFQ056 for the treatment of chorea in Huntington's disease. Mov Disord. 2015 Mar;30(3):427-31. doi: 10.1002/mds.26174. Epub 2015 Feb 17. PMID 25689146